CLINICAL TRIAL: NCT02732431
Title: Obstructive Sleep Apnea Screening and Down Syndrome in Childhood : the Reliability of the Clinical Examination
Brief Title: Obstructive Sleep Apnea and Down Syndrome: Clinical Examination Issue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-HPNCL-06
Record Dates: First submitted 2016-03-22; First posted 2016-04-08 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- trisomy 21 (Other): Parents will complete two sleep symptom questionnaires (PSQ-SRBD and CSHQ) and children will be evaluated by a paediatric pulmonologist and allergist with skin allergy test. An Ear, Nose and Throat specialist will complete two questionnaires (CAS-15 and SCR) carrying a nasopharyngoscopy. Then, children will perform an overnight polysomnography in the Department of Paediatric Functional Investigations of University Hospital in Nice.
  Interventions: Other: Sleep Symptom

INTERVENTIONS:
Other: Sleep Symptom — Questionnaires, skin allergy test, overnight polysomnography

SUMMARY:
Obstructive sleep apnea (OSA) is a common condition of Down syndrome patients. In pediatric practice, there is no way to determine the children with an increased risk. The aim of the study is to determine the reliability of four questionnaires used in pediatric patients in screening of OSA in Down syndrome children.

Prospective study where patients are evaluated on airway diseases and aeroallergens sensitization with 2 parental surveys (PSQ-SRBD and CSHQ), otolaryngologic problems by completing by the ENT surgeon 2 others surveys (CAS-15 and SCR), and sleep disease with an overnight polysomnography (PSG), in University Hospital in Nice.

DETAILED DESCRIPTION:
Introduction: Children with Down syndrome (DS) commonly have obstructive sleep apnea (OSA) though undervalued by parents and physicians. Several sleep questionnaires are used in paediatric patients to detect high risk children who have OSA, but not really appropriate for DS patients. The aim of the study is to determine the reliability of four questionnaires used in paediatric patients (PSQ-SRBD: Pediatric Sleep Questionnaire-Sleep-Related Breathing Disorder, CSHQ: Children's Sleep Habits Questionnaire, CAS-15: Clinical Assessment Score-15 and SCR: Sleep Clinical Record) in screening of OSA in DS population.

Study design: Prospective study concerning children with Down syndrome (age 1-18y). Parents will complete two sleep symptom questionnaires (PSQ-SRBD and CSHQ) and children will be evaluated by a paediatric pulmonologist and allergist with skin allergy test. An Ear, Nose and Throat specialist will complete two questionnaires (CAS-15 and SCR) carrying a nasopharyngoscopy. Then, children will perform an overnight polysomnography in the Department of Paediatric Functional Investigations of University Hospital in Nice.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18 years
* Down syndrome with cytogenetic diagnosis
* State health cover
* Consent of legal representative and/or patient

Exclusion Criteria:

* Polysomnography with correct results during the 12 months before

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
determine the reliability of the Sensitivity of four questionnaires used in paediatric patients in screening of OSA in DS population | At the inclusion
  Sensitivity each survey (PSQ-SRBD, CSHQ, CAS-15, SCR) depending on the obstructive apnea-hypopnea index in the group if children who have an OSA syndrome.

SECONDARY OUTCOMES:
determine the reliability of the specificity of four questionnaires used in paediatric patients in screening of OSA in DS population | At the inclusion
  specificity of each survey (PSQ-SRBD, CSHQ, CAS-15, SCR) depending on the obstructive apnea-hypopnea index in the group if children who have an OSA syndrome.
determine the reliability of positive predictive value of four questionnaires used in paediatric patients in screening of OSA in DS population | At the inclusion
  positive predictive value of each survey (PSQ-SRBD, CSHQ, CAS-15, SCR) depending on the obstructive apnea-hypopnea index in the group if children who have an OSA syndrome.
determine the reliability of negative predictive value of four questionnaires used in paediatric patients in screening of OSA in DS population | At the inclusion
  negative predictive value of each survey (PSQ-SRBD, CSHQ, CAS-15, SCR) depending on the obstructive apnea-hypopnea index in the group if children who have an OSA syndrome.
determine the reliability of positive likelihood ratio of four questionnaires used in paediatric patients in screening of OSA in DS population | At the inclusion
  positive likelihood of each survey (PSQ-SRBD, CSHQ, CAS-15, SCR) depending on the obstructive apnea-hypopnea index in the group if children who have an OSA syndrome.
determine the reliability of negative likelihood ratio of four questionnaires used in paediatric patients in screening of OSA in DS population | At the inclusion
  negative likelihood ratio of each survey (PSQ-SRBD, CSHQ, CAS-15, SCR) depending on the obstructive apnea-hypopnea index in the group if children who have an OSA syndrome.
determine the reliability of area under a receiver operating characteristic (ROC) curve of four questionnaires used in paediatric patients in screening of OSA in DS population | At the inclusion
  area under a receiver operating characteristic (ROC) curve of each survey (PSQ-SRBD, CSHQ, CAS-15, SCR) depending on the obstructive apnea-hypopnea index in the group if children who have an OSA syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: lisa CHAMI, MD, Principal Investigator — Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- CHU de Nice, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: No